CLINICAL TRIAL: NCT03231293
Title: A Multicenter Longitudinal Observational Study to Assess the Effectiveness of Fimasartan-based Antihypertensive Treatment and Prognosis in Post-Acute Phase of Ischemic Stroke or Transient Ischemic Attack
Brief Title: Fimasartan Blood Pressure Lowering After Acute Stroke
Acronym: FABULOUS
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-FMS-OS-401
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Hypertension; Ischemic Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Hypertension; Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This study evaluates the effectiveness of fimasartan-based antihypertensive treatment and prognosis in post-acute phase of ischemic stroke or transient ischemic attack patients. All participants will receive fimasartan, and the investigators will follow them up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke or transient ischemic attack occurs after 7 days to 3 months.
* Mean blood pressure measured 3 times at the first visit (Visit 1) should be over 140 mmHg for systolic blood pressure or 90 mmHg for diastolic blood pressure
* Suitable for administration of fimasartan
* The life expectancy should be over 6 months.

Exclusion Criteria:

* Patients already treated with antihypertensive medications
* Hemorrhagic stroke patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1,032 subjects of post-acute phase of ischemic stroke or transient ischemic attack patients
Sampling Method: Non-Probability Sample
Enrollment: 1035 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
BP | 24 weeks
  Blood pressure control rate(<140/90 mmHg)

SECONDARY OUTCOMES:
BP | 4, 12 weeks
  Blood pressure control rate(<140/90 mmHg)
BP | 4, 12, 24 weeks
  Blood pressure changes
mRS | 4, 12, 24 weeks
  mRS changes
Fimasartan-based treatment | 24 weeks
  Fimasartan-based treatment modalities
Fimasartan starting point | 24 weeks
  Fimasartan starting point after stroke
Stroke recurrence | 24 weeks
  Rate of stroke recurrence
Cardiovascular events | 24 weeks
  Incidence of cardiovascular events
Mortality rates from cardiovascular disease | 24 weeks
  Mortality rates from cardiovascular disease
Mortality rates of any cause | 24 weeks
  Mortality rates of any cause
Adverse events | 24 weeks
  Adverse events related to antihypertensive treatments

CONTACTS AND LOCATIONS:
Overall Officials: Myung Sook Hong, Study Director — Boryung Pharmaceutical Co., Ltd
Locations (27):
- South Korea (27):
  - Korea University Ansan Hospital, Ansan
  - Hallym University Medical Center, Anyang
  - Dong-A University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Daejeon Eulji Medical Center, Daejeon
  - Inje University Ilsan Paik Hospital, Goyang
  - Myongji Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Ewha Womans University Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Kyunghee University Medical Center, Seoul
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Hong KS, Kwon SU, Park JH, Cha JK, Jung JM, Kim YJ, Lee KB, Sohn SI, Lee YS, Rha JH, Kwon JH, Han SW, Kim BJ, Koo J, Choi JC, Sung SM, Lee SJ, Park MS, Ahn SH, Bang OY, Hwang YH, Nam HS, Park JM, Bae HJ, Kim EG, Lee KY, Oh MS. Fimasartan-Based Blood Pressure Control after Acute Cerebral Ischemia: The Fimasartan-Based Blood Pressure Control after Acute Cerebral Ischemia Study. J Clin Neurol. 2021 Jul;17(3):344-353. doi: 10.3988/jcn.2021.17.3.344. PMID 34184441